CLINICAL TRIAL: NCT03863938
Title: A Randomized, Open-label, Single-dose Phase 1 Clinical Trial to Compare the Effect of Timing of Food on the Pharmacokinetics and Pharmacodynamics of K-CAB (Tegoprazan) in Healthy Male Subjects
Brief Title: Food-Effect on PK and PD of Single Oral Dose of Tegoprazan in Healthy Male Subjects
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: HK inno.N Corporation (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: CJ_APA_112
Record Dates: First submitted 2019-02-28; First posted 2019-03-05 (Actual); Last update posted 2019-08-22 (Actual); Status verified 2019-08

CONDITIONS: Healthy
MeSH Terms: interventions — tegoprazan; Tablets

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Tegoprazan 50mg under fasting condition (Experimental): Treatment A: single oral administration of Tegoprazan 50mg tablet under fasting condition once a day
  Interventions: Drug: Tegoprazan 50mg
- Tegoprazan 50mg before the meal (Experimental): Treatment B: single oral administration of Tegoprazan 50mg tablet before the meal once a day
  Interventions: Drug: Tegoprazan 50mg
- Tegoprazan 50mg after the meal (Experimental): Treatment C: single oral administration of Tegoprazan 50mg tablet after the meal once a day
  Interventions: Drug: Tegoprazan 50mg

INTERVENTIONS:
Drug: Tegoprazan 50mg — K-CAB
  Other Names: Tegoprazan 50mg tablet

SUMMARY:
This study aims to evaluate the food-effect of tegoprazan 50mg on the pharmacokinetics and pharmacodynamics in healthy H. pylori negative male volunteers

DETAILED DESCRIPTION:
Primary Outcome Measure:

1. AUClast and Cmax of tegaprazan
2. Gastric pH

ELIGIBILITY:
Inclusion Criteria:

* Healthy adult males aged ≥ 19 years and ≤ 50 years
* Body weight of ≥ 55.0 kg and ≤ 90.0 kg, with body mass index (BMI) of ≥ 18.0 kg/m2 and ≤ 27.0 kg/m2 at the time of screening
* Helicobacter pylori negative

Exclusion Criteria:

* Presence or history of clinically significant diseases
* Presence or history of gastrointestinal disorder (gastric ulcer, GERD, Crohn's disease, etc.)
* Hypersensitivity to drugs containing study drug or proton pump inhibitor and other drugs (aspirin, antibiotics, etc.) or history of clinically significant hypersensitivity
* Serologic test positive
* Abnormal obstacle to insertion and maintenance of pH meter catheter
* History of drug abuse
* Excessive caffeine intake or persistent alcohol intake
* Not use of a medically acceptable method of contraception

Ages: 19 Years to 50 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 12 (Actual)
Dates: Start 2019-03-27 (Actual); Primary Completion 2019-04-26 (Actual); Study Completion 2019-06-25 (Actual)

PRIMARY OUTCOMES:
AUClast of tegaprazan | Pre-dose(0 hour) and up to 48 hours in each period
  Area under the plasma concentration versus time curve of tegoprazan
Cmax of tegaprazan | Pre-dose(0 hour) and up to 48 hours in each period
  Peak Plasma Concentration of tegoprazan
Gastric pH | Pre-dose(0 hour) up to 24 hours after Investigational product administration in each period
  Gastric pH

CONTACTS AND LOCATIONS:
Overall Officials: In-Jin Jang, MD, PhD, Principal Investigator — Seoul National University Hospital, Dept. of Clinical Pharmacology
Locations (1):
- Seoul National University Hospital, Clinical Trial Center, Seoul, South Korea